CLINICAL TRIAL: NCT05656950
Title: Assessment of Oral Health Status of Patients in Pediatric Intensive Care Units
Acronym: PICU
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, RAMAZANBOZKURT, Research Assistant, Sakarya University
Other Study IDs: oral assessment pediatric
Record Dates: First submitted 2022-12-10; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Assessment of Oral Health Status of Patients in Pediatric Intensive Care Units
Keywords: Pediatric intensive care unit; Oral health; Oral care; Oral health assessment
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed: Oral health of the patient was evaluated by the researcher using a flashlight, tongue depressor and Oral Evaluation Guide. Patient's age, gender, day of hospitalization in pediatric intensive care units, medical diagnosis/diagnoses, presence of chronic disease, state of consciousness, body temperature, oral care application method, oral care application frequency, oral care product used, amount taken/extracted, drugs used, albumin and haemoglobin data on values were obtained from the observation form of the patient.
  Interventions: Procedure: Assessment

INTERVENTIONS:
Procedure: Assessment — Oral health of the patient was evaluated by the researcher using a flashlight, tongue depressor and Oral Evaluation Guide.

SUMMARY:
The research is a descriptive study designed to evaluate the oral health status of hospitalized children in pediatric intensive care units. The research was conducted between June 2021 and September 2021 in pediatric intensive care units in Izmir province. The patients were included in the study by using the cluster sampling method in the selection of the sample (n=88). Patient Identification Information Form and Oral Assessment Guide (OAG) were used for oral health assessment of patients. It was taken written consents from the hospitals where the research was carried out and from the relatives of the patients

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the PICU
* Parent's consent to participate in the study

Exclusion Criteria:

* Applying non-invasive ventilation therapy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Under 18 ages
Study Population: Under 18 years old patients who are therapy in PICU
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Assessing oral status of children in pediatric intensive care unit | 3 months
  Oral health of the patient was evaluated using a flashlight and tongue depressor

CONTACTS AND LOCATIONS:
Locations (1):
- Ramazan Bozkurt, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akkaş, I., Toptaş, O., ve Özan, F. (2014). Ağız kuruluğu. Acta Odontol Turc, 31(1), 54-60.
- [Background] Barbosa de Castro Piau CG, Azevedo TD, de Castro Piau AG, Miranda AF, Pinheiro JA, Bezerra AC. Oral Microbial Colonization in Pediatric Intensive Care Unit Patients. J Dent Child (Chic). 2016;83(2):53-9. PMID 27620514
- [Background] Labeau SO, Blot SI. Toothbrushing for preventing ventilator-associated pneumonia. Crit Care. 2013 Mar 5;17(2):417. doi: 10.1186/cc12511. No abstract available. PMID 23462424
- [Background] Maeda K, Akagi J. Oral care may reduce pneumonia in the tube-fed elderly: a preliminary study. Dysphagia. 2014 Oct;29(5):616-21. doi: 10.1007/s00455-014-9553-6. Epub 2014 Jul 18. PMID 25034303
- [Background] Nederfors T. Xerostomia and hyposalivation. Adv Dent Res. 2000 Dec;14:48-56. doi: 10.1177/08959374000140010701. PMID 11842923
- [Background] Hocherman S, Yirmiya R. Neuronal activity in the medial geniculate nucleus and in the auditory cortex of the rhesus monkey reflects signal anticipation. Brain. 1990 Dec;113 ( Pt 6):1707-20. doi: 10.1093/brain/113.6.1707. PMID 2276042
- [Background] Walls AW, Steele JG. The relationship between oral health and nutrition in older people. Mech Ageing Dev. 2004 Dec;125(12):853-7. doi: 10.1016/j.mad.2004.07.011. PMID 15563930
- [Result] Abidia RF. Oral care in the intensive care unit: a review. J Contemp Dent Pract. 2007 Jan 1;8(1):76-82. PMID 17211508
- [Result] Ames NJ, Sulima P, Yates JM, McCullagh L, Gollins SL, Soeken K, Wallen GR. Effects of systematic oral care in critically ill patients: a multicenter study. Am J Crit Care. 2011 Sep;20(5):e103-14. doi: 10.4037/ajcc2011359. PMID 21885453
- [Result] Berry AM, Davidson PM. Beyond comfort: oral hygiene as a critical nursing activity in the intensive care unit. Intensive Crit Care Nurs. 2006 Dec;22(6):318-28. doi: 10.1016/j.iccn.2006.04.003. Epub 2006 Jun 27. PMID 16806933
- [Result] Berry AM, Davidson PM, Nicholson L, Pasqualotto C, Rolls K. Consensus based clinical guideline for oral hygiene in the critically ill. Intensive Crit Care Nurs. 2011 Aug;27(4):180-5. doi: 10.1016/j.iccn.2011.04.005. PMID 21684164
- [Result] Celik GG, Eser I. Examination of intensive care unit patients' oral health. Int J Nurs Pract. 2017 Dec;23(6). doi: 10.1111/ijn.12592. Epub 2017 Sep 28. PMID 28960619
- [Result] Chang I, Schibler A. Ventilator Associated Pneumonia in Children. Paediatr Respir Rev. 2016 Sep;20:10-16. doi: 10.1016/j.prrv.2015.09.005. Epub 2015 Sep 25. PMID 26527358
- [Result] Cheng KK. Children's acceptance and tolerance of chlorhexidine and benzydamine oral rinses in the treatment of chemotherapy-induced oropharyngeal mucositis. Eur J Oncol Nurs. 2004 Dec;8(4):341-9. doi: 10.1016/j.ejon.2004.04.002. PMID 15550364
- [Result] Çiftcioğlu, Ş., ve Efe, E. (2017). Validity and reliability of the oral assessment guide for children and young people receiving chemotherapy. Turk Onkoloji Dergisi, 32(4), 133-140. https://doi.org/10.5505/tjo.2017.1671
- [Result] Collins T, Plowright C, Gibson V, Stayt L, Clarke S, Caisley J, Watkins CH, Hodges E, Leaver G, Leyland S, McCready P, Millin S, Platten J, Scallon M, Tipene P, Wilcox G. British Association of Critical Care Nurses: Evidence-based consensus paper for oral care within adult critical care units. Nurs Crit Care. 2021 Jul;26(4):224-233. doi: 10.1111/nicc.12570. Epub 2020 Oct 29. PMID 33124119
- [Result] Cutler CJ, Davis N. Improving oral care in patients receiving mechanical ventilation. Am J Crit Care. 2005 Sep;14(5):389-94. PMID 16120890
- [Result] Dogu Kokcu O, Terzi B. Development of an intensive care oral care frequency assessment scale. Nurs Crit Care. 2022 Sep;27(5):667-675. doi: 10.1111/nicc.12529. Epub 2020 Jul 6. PMID 32633044
- [Result] Ettinger RL. Review: xerostomia: a symptom which acts like a disease. Age Ageing. 1996 Sep;25(5):409-12. doi: 10.1093/ageing/25.5.409. PMID 8921150
- [Result] Franklin D, Senior N, James I, Roberts G. Oral health status of children in a Paediatric Intensive Care Unit. Intensive Care Med. 2000 Mar;26(3):319-24. doi: 10.1007/s001340051156. PMID 10823389
- [Result] DeKeyser Ganz F, Fink NF, Raanan O, Asher M, Bruttin M, Nun MB, Benbinishty J. ICU nurses' oral-care practices and the current best evidence. J Nurs Scholarsh. 2009;41(2):132-8. doi: 10.1111/j.1547-5069.2009.01264.x. PMID 19538697
- [Result] Glenny AM, Gibson F, Auld E, Coulson S, Clarkson JE, Craig JV, Eden OB, Khalid T, Worthington HV, Pizer B; Children's Cancer and Leukaemia Group (CCLG)/Paediatric Oncology Nurses Forum's (CCLG-PONF) Mouth Care Group. The development of evidence-based guidelines on mouth care for children, teenagers and young adults treated for cancer. Eur J Cancer. 2010 May;46(8):1399-412. doi: 10.1016/j.ejca.2010.01.023. Epub 2010 Mar 11. PMID 20227272
- [Result] Gomes GF, Pisani JC, Macedo ED, Campos AC. The nasogastric feeding tube as a risk factor for aspiration and aspiration pneumonia. Curr Opin Clin Nutr Metab Care. 2003 May;6(3):327-33. doi: 10.1097/01.mco.0000068970.34812.8b. PMID 12690267
- [Result] Grap MJ, Munro CL, Ashtiani B, Bryant S. Oral care interventions in critical care: frequency and documentation. Am J Crit Care. 2003 Mar;12(2):113-8; discussion 119. PMID 12625169
- [Result] Grap MJ, Munro CL, Elswick RK Jr, Sessler CN, Ward KR. Duration of action of a single, early oral application of chlorhexidine on oral microbial flora in mechanically ventilated patients: a pilot study. Heart Lung. 2004 Mar-Apr;33(2):83-91. doi: 10.1016/j.hrtlng.2003.12.004. PMID 15024373
- [Result] Grinspun, D. (2008). Oral Health : Nursing Assessment and Interventions. Nursing Best Practice Guideline, December, 99. www.rnao.org/bestpractices
- [Result] Gunes Z, Denat Y, Muezzinoglu M, Sen S, Yilmaz S, Atli E. The risk factors effecting the dry mouth in inpatients in Hospital in west Anatolia. J Clin Nurs. 2012 Feb;21(3-4):408-14. doi: 10.1111/j.1365-2702.2011.03898.x. Epub 2011 Nov 18. PMID 22098453
- [Result] Hanneman SK, Gusick GM. Frequency of oral care and positioning of patients in critical care: a replication study. Am J Crit Care. 2005 Sep;14(5):378-86; quiz 387. PMID 16120889
- [Result] Hanonu S, Karadag A. A Prospective, Descriptive Study to Determine the Rate and Characteristics of and Risk Factors for the Development of Medical Device-related Pressure Ulcers in Intensive Care Units. Ostomy Wound Manage. 2016 Feb;62(2):12-22. PMID 26901386
- [Result] Cooper VB, Haut C. Preventing ventilator-associated pneumonia in children: an evidence-based protocol. Crit Care Nurse. 2013 Jun;33(3):21-9; quiz 30. doi: 10.4037/ccn2013204. PMID 23727849
- [Result] Houston S, Hougland P, Anderson JJ, LaRocco M, Kennedy V, Gentry LO. Effectiveness of 0.12% chlorhexidine gluconate oral rinse in reducing prevalence of nosocomial pneumonia in patients undergoing heart surgery. Am J Crit Care. 2002 Nov;11(6):567-70. PMID 12425407
- [Result] Human, L., ve Bell, J. (2007). Oral hygiene care in critically ill patients. Southern African Journal of Critical Care, 23(2), 61-65. https://doi.org/10.7196/SAJCC.24
- [Result] Jablonski S. Oral rehydration of the pediatric patient with mild to moderate dehydration. J Emerg Nurs. 2012 Mar;38(2):185-7; quiz 201. doi: 10.1016/j.jen.2011.12.001. Epub 2012 Jan 14. No abstract available. PMID 22245399
- [Result] Johnstone L, Spence D, Koziol-McClain J. Oral hygiene care in the pediatric intensive care unit: practice recommendations. Pediatr Nurs. 2010 Mar-Apr;36(2):85-96; quiz 97. PMID 20476510
- [Result] McConnell ES, Lekan D, Hebert C, Leatherwood L. Academic-practice partnerships to promote evidence-based practice in long-term care: oral hygiene care practices as an exemplar. Nurs Outlook. 2007 Mar-Apr;55(2):95-105. doi: 10.1016/j.outlook.2006.12.003. PMID 17386313
- [Result] McNeill HE. Biting back at poor oral hygiene. Intensive Crit Care Nurs. 2000 Dec;16(6):367-72. doi: 10.1054/iccn.2000.1531. PMID 11091468
- [Result] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Result] Mohammed, H. M., ve Hassan, M. S. (2015). Endotracheal tube securements: Effectiveness of three techniques among orally intubated patients. Egyptian Journal of Chest Diseases and Tuberculosis, 64(1), 183-196. https://doi.org/10.1016/j.ejcdt.2014.09.006
- [Result] Munro CL, Grap MJ. Oral health and care in the intensive care unit: state of the science. Am J Crit Care. 2004 Jan;13(1):25-33; discussion 34. PMID 14735645
- [Result] Munro CL, Grap MJ, Jablonski R, Boyle A. Oral health measurement in nursing research: state of the science. Biol Res Nurs. 2006 Jul;8(1):35-42. doi: 10.1177/1099800406289343. PMID 16766627
- [Result] O'Reilly M. Oral care of the critically ill: a review of the literature and guidelines for practice. Aust Crit Care. 2003 Aug;16(3):101-10. doi: 10.1016/s1036-7314(03)80007-3. PMID 14533214
- [Result] Prasanthi B, Kannan N, Patil R. Effect of Diuretics on Salivary Flow, Composition and Oral Health Status: A Clinico-biochemical Study. Ann Med Health Sci Res. 2014 Jul;4(4):549-53. doi: 10.4103/2141-9248.139311. PMID 25221702
- [Result] Pedreira ML, Kusahara DM, de Carvalho WB, Nunez SC, Peterlini MA. Oral care interventions and oropharyngeal colonization in children receiving mechanical ventilation. Am J Crit Care. 2009 Jul;18(4):319-28; quiz 329. doi: 10.4037/ajcc2009121. PMID 19556410
- [Result] Prendergast, V. Safety and Efficacy of Oral Care for Intubated Neuroscience Intensive Care Unit Patients (Issue 37). 2012. Lund University.
- [Result] Prendergast V, Kleiman C, King M. The Bedside Oral Exam and the Barrow Oral Care Protocol: translating evidence-based oral care into practice. Intensive Crit Care Nurs. 2013 Oct;29(5):282-90. doi: 10.1016/j.iccn.2013.04.001. Epub 2013 May 20. PMID 23702324
- [Result] Rello J, Koulenti D, Blot S, Sierra R, Diaz E, De Waele JJ, Macor A, Agbaht K, Rodriguez A. Oral care practices in intensive care units: a survey of 59 European ICUs. Intensive Care Med. 2007 Jun;33(6):1066-70. doi: 10.1007/s00134-007-0605-3. Epub 2007 Mar 24. PMID 17384927
- [Result] Schunemann, F. H., Canani, S. H., ve Marín, C. (2017). Oral evaluation of children and adolescents in intensive care unit. Rsbo, 14(3), 135-141. https://doi.org/10.21726/rsbo.v1i3.482
- [Result] Sreenivasan VPD, Ganganna A, Rajashekaraiah PB. Awareness among intensive care nurses regarding oral care in critically ill patients. J Indian Soc Periodontol. 2018 Nov-Dec;22(6):541-545. doi: 10.4103/jisp.jisp_30_18. PMID 30631234
- [Result] Turk G, Kocacal Guler E, Eser I, Khorshid L. Oral care practices of intensive care nurses: a descriptive study. Int J Nurs Pract. 2012 Aug;18(4):347-53. doi: 10.1111/j.1440-172X.2012.02045.x. PMID 22845634
- [Result] Ullman A, Long D, Lewis P. The oral health of critically ill children: an observational cohort study. J Clin Nurs. 2011 Nov;20(21-22):3070-80. doi: 10.1111/j.1365-2702.2011.03797.x. Epub 2011 Aug 1. PMID 21801254
- [Result] Velazco CS, Zurakowski D, Fullerton BS, Bechard LJ, Jaksic T, Mehta NM. Nutrient delivery in mechanically ventilated surgical patients in the pediatric critical care unit. J Pediatr Surg. 2017 Jan;52(1):145-148. doi: 10.1016/j.jpedsurg.2016.10.041. Epub 2016 Oct 28. PMID 27856012
- [Result] Yildiz M, Durna Z, Akin S. Assessment of oral care needs of patients treated at the intensive care unit. J Clin Nurs. 2013 Oct;22(19-20):2734-47. doi: 10.1111/jocn.12035. Epub 2013 Mar 27. PMID 23534462
- [Derived] Bozkurt R, Eser I. Assessment of the Oral Health Status of Patients Admitted to Pediatric Intensive Care Units: A Cross-Sectional Study. Dimens Crit Care Nurs. 2024 Mar-Apr 01;43(2):53-60. doi: 10.1097/DCC.0000000000000625. PMID 38271308